CLINICAL TRIAL: NCT07260838
Title: The Effect of Showing Fetal Images to High-Risk Pregnant Women on Pregnancy Stress and Sleep Quality
Brief Title: The Effect of Showing Fetal Images to High-Risk Pregnant Women on Stress and Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melike Nur SÖNMEZ (Other)
Responsible Party: Sponsor-Investigator, Melike Nur SÖNMEZ, Master's Student Researcher, Cukurova University
Organization: Cukurova University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 147-67/06.09.2024
Record Dates: First submitted 2025-11-16; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy, High-Risk
Keywords: Risky Pregnancy; Fetal Imaging; Pregnancy Stress; Sleep Quality; Nursing
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Fetal images were shown.) (Experimental): The video containing fetal images will be shown to participants in the intervention group. Support will be obtained from the clinical doctor in preparing this video. At the clinic, each pregnant woman will have a video of her own fetus recorded using an ultrasound device in the examination room, and each pregnant woman will watch the video containing her own fetal images.
  Interventions: Other: Showing fetal images
- Control Group (No Intervention): The researcher will not intervene with the pregnant women in the control group.

INTERVENTIONS:
Other: Showing fetal images — High-risk pregnant women in the intervention group were shown fetal images three times a day for two days.
  Arms: Intervention Group (Fetal images were shown.)

SUMMARY:
The study will be conducted to determine the effect of showing fetal images to high-risk pregnant women on pregnancy stress and sleep quality.

The study was conducted at Adana City Training and Research Hospital between November 2024 and May 2025 using a randomized controlled, interventional design. The sample of the study consisted of 35 intervention and 35 control group participants, totaling 70 individuals. Data were collected using the Personal Information Form, the Pregnancy Stress Rating Scale (PSRS-36) and the Richard-Campbell Sleep Scale. The intervention group was shown fetal images three times a day for two days; the control group received no intervention. The collected data were analyzed by comparing the pre-test and post-test scores. The data obtained from the study will be evaluated using SPSS IBM 24.0 package program in computer environment.

Research Hypotheses:

In the intervention and control groups; H0-1: Showing fetal images to high-risk pregnant women has no effect on pregnancy stress.

H0-2: Showing fetal images to high-risk pregnant women has no effect on sleep quality.

H1-1: Showing fetal images to high-risk pregnant women has an effect on pregnancy stress.

H1-2: Showing fetal images to high-risk pregnant women has an effect on sleep quality.

DETAILED DESCRIPTION:
This study was supported by the Scientific Research Projects Coordination Unit (BAP) of Çukurova University, Project Code: [TYL-2025-17328].

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 45
* Having an educational background of elementary school or higher
* Being at least 20 weeks pregnant
* Having a planned hospital stay of at least 3 days
* Being hospitalized for the first time during pregnancy
* Being able to speak Turkish
* Being able to communicate verbally

Exclusion Criteria:

* Having previously participated in the practice of viewing fetal images
* Diagnosis of mental illness
* Becoming pregnant through infertility treatment
* Presence of visual/hearing impairment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study only covers women with high-risk pregnancies.
Enrollment: 70 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-05-17 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
The effect of showing fetal images to high-risk pregnant women on pregnancy stress | Three times a day for two days
  Pregnancy Stress Rating Scale; The scale is a 5-Likert type. The degree of anxiety, distress, and worry experienced by pregnant women is rated as "definitely no," "mild," "moderate," "severe," or "very severe," and scores range from 0 to 4. Perceived stress levels during pregnancy range from a minimum of 0 to a maximum of 144 points. Higher scores on the scale indicate increased stress.
The effect of showing fetal images to high-risk pregnant women on sleep quality | Three times a day for two days
  Richard-Campbell Sleep Scale; The scale consists of 6 items. Each item is rated on a visual analog scale ranging from 0 to 100. A score between "0-25" on the scale indicates very poor sleep, while a score between "76-100" indicates very good sleep. The total scale score is evaluated based on 5 items; the 6th item, which assesses the noise level in the environment, is excluded from the total score evaluation. As the scale score increases, patients' sleep quality improves.

CONTACTS AND LOCATIONS:
Overall Officials: EVŞEN NAZİK, Professor, Study Director — Çukurova University Faculty of Health Sciences
Locations (1):
- Adana City Training and Research Hospital, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
To protect participant confidentiality and ensure ethical compliance, individual participant data will not be shared.